CLINICAL TRIAL: NCT00066937
Title: Pain Management in Temporomandibular Joint Disorders
Brief Title: Comparison of Psychological and Pharmacological Treatments for Pain Due to Temporomandibular Joint Disorder (TMD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPN 00-03-21-02; R01DE013906 (NIH)
Record Dates: First submitted 2003-08-07; First posted 2003-08-08 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-07

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Nortriptyline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Nortriptyline Oral Capsule/CBT (Experimental): Nortriptyline taken at bedtime titrated to a dose up to 150 mg. Study participants also receive 6 sessions of CBT.
  Interventions: Drug: Nortriptyline Oral Capsule; Behavioral: CBT
- Benztropine Oral Product/CBT (Experimental): Benztropine will be titrated up from .125 mg qhs to a maximum dose of .750 mg qhs based on treatment response and side effect profile. Study participants also receive 6 sessions of CBT.
  Interventions: Drug: Benztropine Oral Product; Behavioral: CBT
- Nortriptyline Oral Capsule/Disease MGT (Experimental): Nortriptyline taken at bedtime titrated to a dose up to 150 mg. Study participants also receive 6 sessions of TMD disease management.
  Interventions: Drug: Nortriptyline Oral Capsule; Behavioral: Disease MGT
- Benztropine Oral Product/Disease MGT (Active Comparator): Benztropine will be titrated up from .125 mg qhs to a maximum dose of .750 mg qhs based on treatment response and side effect profile. Study participants also receive 6 sessions of TMD disease management.
  Interventions: Drug: Benztropine Oral Product; Behavioral: Disease MGT

INTERVENTIONS:
Drug: Nortriptyline Oral Capsule — Nortriptyline will be titrated up from 25 mg qhs to a maximum dose of 150 mg qhs based on treatment response and side effect profile.
  Arms: Nortriptyline Oral Capsule/CBT; Nortriptyline Oral Capsule/Disease MGT
Drug: Benztropine Oral Product — Benztropine will be titrated up from .125 mg qhs to a maximum dose of .750 mg qhs based on treatment response and side effect profile.
  Arms: Benztropine Oral Product/CBT; Benztropine Oral Product/Disease MGT
Behavioral: CBT — Six in-person, individual sessions of cognitive-behavioral therapy for pain management include relaxation training, pain coping skills training, cognitive therapy for negative and dysfunctional thoughts, and diaries for monitoring relaxation, goals, and negative thinking.
  Arms: Benztropine Oral Product/CBT; Nortriptyline Oral Capsule/CBT
Behavioral: Disease MGT — Six in-person, individual sessions of temporomandibular joint disorder (TMD) disease management (MGT) that include information about the jaw and good oral habits, diet, sleep, and general stress management.
  Arms: Benztropine Oral Product/Disease MGT; Nortriptyline Oral Capsule/Disease MGT

SUMMARY:
The purpose of this study is to determine whether the combination of cognitive-behavioral treatment and nortriptyline are more effective than each treatment alone in reducing the pain and disability associated with TMD.

DETAILED DESCRIPTION:
This is a randomized, controlled trial evaluating pharmacological (nortriptyline vs. active placebo - benztropine) and psychological (cognitive-behavioral therapy vs. disease education) treatments for pain and disability due to temporomandibular joint disorder (TMD). Patients 18 to 65 years old meeting RDC criteria for TMD and other eligibility criteria complete a 3-week baseline monitoring phase prior to randomization. Active treatment consists of weekly visits for 8 week, then maintenance treatment for 6 months. Outcome measures include pain, physical and psychosocial function and are assessed at post-treatment, 3-months, and 6-months

ELIGIBILITY:
Inclusion:

* Age >= 18 and <= 65
* Pain >= 3 months duration due to temporomandibular joint disorder
* Pain due to TMD is primary if other pain conditions present

Exclusion:

* Continuous, chronic painful non-reducing disc displacement of TMJ and patient can't open mouth
* Unstable or acute severe pain from another pain condition
* Patient is pregnant
* Presence of a medical condition that contraindicates nortriptyline: angle-closure glaucoma,symptomatic orthosis
* EKG: first degree heart block or QTc > 450 msec
* Unstable angina or a history of a myocardial infarction within the past 3 months
* Current treatment with an antidepressant which cannot be withdrawn
* Current use of a medication that interacts with nortriptyline to raise blood levels, such as selective serotonin reuptake inhibitors (e.g.,paroxetine), systemic anti-fungal agents (fluconazole), antiarrhythmics (e.g., quinidine), antipsychotics (e.g., haloperidol), and antibiotics (e.g., erythromycin).
* Presence of dementia, psychosis or other disorder of cognition that impairs ability to participate in minimal contact intervention
* Beck Depression Inventory (BDI) score >= 35 OR BDI Item #9 (suicide item) is scored > 1
* Patient has a terminal illness with a life expectancy of less than six months
* History of arthrotomy of temporomandibular joint
* History of allergic reaction to nortriptyline or benztropine
* History of a therapeutic trial with nortriptyline (dose >= 100 mg for at least 3 weeks)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2002-11; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Haythornthwaite, Ph.D, Principal Investigator — Johns Hopkins University
Locations (1):
- University of Maryland, Dental School, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Treatment Phase
Arm/Group | Nortriptyline Oral Capsule/CBT | Benztropine Oral Product/CBT | Nortriptyline Oral Capsule/Disease MGT | Benztropine Oral Product/Disease MGT
Started | 41 | 38 | 37 | 24
Completed | 38 | 33 | 26 | 19
Not Completed | 3 | 5 | 11 | 5
Period: 3 Month Follow-up
Arm/Group | Nortriptyline Oral Capsule/CBT | Benztropine Oral Product/CBT | Nortriptyline Oral Capsule/Disease MGT | Benztropine Oral Product/Disease MGT
Started | 38 | 33 | 26 | 19
Completed | 33 | 32 | 25 | 15
Not Completed | 5 | 1 | 1 | 4
Period: 6 Month Follow-up
Arm/Group | Nortriptyline Oral Capsule/CBT | Benztropine Oral Product/CBT | Nortriptyline Oral Capsule/Disease MGT | Benztropine Oral Product/Disease MGT
Started | 33 | 32 | 25 | 15
Completed | 26 | 29 | 22 | 14
Not Completed | 7 | 3 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nortriptyline Oral Capsule/CBT | Benztropine Oral Product/CBT | Nortriptyline Oral Capsule/Disease MGT | Benztropine Oral Product/Disease MGT | Total
Number analyzed (Participants) | 41 | 38 | 37 | 24 | 140
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.7 (12.0) | 38.4 (12.5) | 37.2 (11.5) | 33.3 (11.3) | 36.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 29 | 28 | 17 | 105
  Male | 10 | 9 | 9 | 7 | 35
Region of Enrollment [Number; unit: participants]
  United States | 41 | 38 | 37 | 24 | 140

OUTCOME MEASURES:

1. Primary Outcome: Average Pain
Description: 0 (no pain) to 10 (pain as bad as could be) rating of average pain during the past week; higher scores indicate greater pain
Time Frame: baseline, post-treatment, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nortriptyline Oral Capsule/CBT | Benztropine Oral Product/CBT | Nortriptyline Oral Capsule/Disease MGT | Benztropine Oral Product/Disease MGT
Number analyzed (Participants) | 38 | 33 | 26 | 19
units on a scale
  baseline | 4.7 (2.2) | 4.4 (2.1) | 4.5 (2.2) | 5.0 (1.8)
  post treatment | 2.8 (2.6) | 2.7 (2.1) | 2.0 (1.4) | 2.8 (2.1)
  3 months | 2.1 (1.6) | 2.4 (2.2) | 2.2 (2.1) | 2.5 (2.1)
  6 months | 2.0 (1.7) | 2.0 (2.1) | 1.4 (1.6) | 2.2 (2.5)
Statistical Analysis 1: Comparison: Nortriptyline Oral Capsule/CBT vs Benztropine Oral Product/CBT vs Nortriptyline Oral Capsule/Disease MGT vs Benztropine Oral Product/Disease MGT; Test type: Other; p < .05, ANOVA; Repeated measures ANOVAs compared baseline to each timepoint

2. Primary Outcome: Change in Pain-related Interference
Description: Multidimensional Pain Inventory: Pain interference subscale score; average score computed from 12 items rated on scale from 0=no interference to 6=extreme interference; higher scores indicate greater pain-related interference
Time Frame: baseline, post-treatment, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Nortriptyline Oral Capsule/CBT | Benztropine Oral Product/CBT | Nortriptyline Oral Capsule/Disease MGT | Benztropine Oral Product/Disease MGT
Number analyzed (Participants) | 38 | 33 | 26 | 19
Change in scores on a scale
  Change in score from baseline to post-treatment | 0.9 (0.9) | 0.5 (0.9) | 0.5 (0.7) | 1.0 (0.9)
  Change in score from baseline to 3 months | 0.8 (0.9) | 0.8 (0.9) | 1.0 (0.9) | 1.1 (1.2)
  Change in score from baseline to 6 months | 0.8 (0.8) | 0.7 (1.2) | 0.7 (0.8) | 0.8 (1.1)
Statistical Analysis 1: Comparison: Nortriptyline Oral Capsule/CBT vs Benztropine Oral Product/CBT vs Nortriptyline Oral Capsule/Disease MGT vs Benztropine Oral Product/Disease MGT; Test type: Other; p < .05, ANOVA; Repeated measures ANOVAs compared baseline scores to each period of follow-up (post-treatment, 3-months, 6 months)

3. Secondary Outcome: Worst Pain
Description: 0 (no pain) to 10 (pain as bad as could be) rating of worst pain during the past week
Time Frame: baseline, post-treatment, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nortriptyline Oral Capsule/CBT | Benztropine Oral Product/CBT | Nortriptyline Oral Capsule/Disease MGT | Benztropine Oral Product/Disease MGT
Number analyzed (Participants) | 38 | 33 | 26 | 19
units on a scale
  baseline | 6.7 (2.3) | 6.1 (2.2) | 6.3 (2.4) | 7.2 (1.9)
  post-treatment | 4.0 (2.9) | 4.1 (2.8) | 3.2 (2.1) | 4.4 (2.6)
  3 months | 3.6 (2.4) | 3.3 (2.3) | 3.4 (2.7) | 4.1 (2.9)
  6 months | 3.3 (2.1) | 3.1 (2.7) | 2.7 (2.2) | 3.4 (2.9)
Statistical Analysis 1: Comparison: Nortriptyline Oral Capsule/CBT vs Benztropine Oral Product/CBT vs Nortriptyline Oral Capsule/Disease MGT vs Benztropine Oral Product/Disease MGT; Test type: Other; p < .05, ANOVA; Repeated measures ANOVAs compared baseline scores to each period of follow-up (post-treatment, 3-months, 6 months)

4. Secondary Outcome: Mental Health as Assessed by the Short Form 36 Healthy Survey
Description: The Mental Health Component score from the Short Form (36) Health Survey, which is a 36-item, patient-reported survey of patient health. The mental health component score is calculated from responses to the general health, mental health, vitality, physical and emotional role limitations, and social functioning subscales, with higher scores indicating better mental health. The scale ranges from zero (equivalent to maximum disability) to 100 (no disability).
Time Frame: baseline, post-treatment, 3 months, 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nortriptyline Oral Capsule/CBT | Benztropine Oral Product/CBT | Nortriptyline Oral Capsule/Disease MGT | Benztropine Oral Product/Disease MGT
Number analyzed (Participants) | 38 | 33 | 26 | 19
units on a scale
  baseline | 50.5 (8.1) | 49.2 (9.3) | 51.2 (8.8) | 48.0 (8.9)
  post-treatment | 50.8 (10.4) | 48.4 (8.1) | 52.6 (10.0) | 53.3 (10.6)
  3 months | 51.5 (8.9) | 50.2 (8.7) | 52.6 (10.0) | 53.8 (10.1)
  6 months | 52.2 (7.8) | 53.3 (12.8) | 52.3 (7.2) | 53.6 (7.3)
Statistical Analysis 1: Comparison: Nortriptyline Oral Capsule/CBT vs Benztropine Oral Product/CBT vs Nortriptyline Oral Capsule/Disease MGT vs Benztropine Oral Product/Disease MGT; Test type: Other; p < .05, ANOVA; Repeated measures ANOVAs compared baseline scores to each period of follow-up (post-treatment, 3-months, 6 months)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected weekly during the treatment phase, then at 3- and 6-months
Arm/Group | Nortriptyline Oral Capsule/CBT | Benztropine Oral Product/CBT | Nortriptyline Oral Capsule/Disease MGT | Benztropine Oral Product/Disease MGT
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/38 | 0/37 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/38 | 0/37 | 0/24
Other Adverse Events (participants affected / at risk) | 32/41 | 24/38 | 21/37 | 15/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nortriptyline Oral Capsule/CBT (N=41) | Benztropine Oral Product/CBT (N=38) | Nortriptyline Oral Capsule/Disease MGT (N=37) | Benztropine Oral Product/Disease MGT (N=24)
drymouth (General disorders) | 20 | 14 | 13 | 9
sedation (Nervous system disorders) | 7 | 8 | 7 | 3
constipation (Gastrointestinal disorders) | 10 | 7 | 9 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No